CLINICAL TRIAL: NCT06343363
Title: Early Discharge After Mitral and Tricuspid Edge-to-edge Repair: an Assessment of Feasibility and Safety
Acronym: EARLY-Edge
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Sam Dawkins, Primary Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: 318352
Record Dates: First submitted 2023-10-29; First posted 2024-04-02 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Mitral Regurgitation; Tricuspid Regurgitation; Mitral Repair; Heart Failure
Keywords: transcatheter edge-to-edge repair; mitral TEER; mitral regurgitation; tricuspid regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency; Tricuspid Valve Insufficiency; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients treated with either mitral TEER, tricuspid TEER or both: Patients treated with either mitral TEER, tricuspid TEER or both, at John Radcliffe Hospital, Oxford
  Interventions: Behavioral: Early discharge protocol

INTERVENTIONS:
Behavioral: Early discharge protocol — Patients admitted for transcatheter edge-to-edge repair to either mitral or tricuspid valve and then discharged within 36 hours

SUMMARY:
Mitral regurgitation (MR) and tricuspid regurgitation (TR) are common causes of breathlessness, fluid retention and other heart failure symptoms, which lead to reduced quality of life and frequent hospitalisation. These conditions are particularly prevalent in older adults with many of these patients being at high risk for surgical intervention due to frailty and comorbidities, leaving them with few treatment alternatives.

Transcatheter edge-to-edge repair (TEER) procedures have increasingly been used to improve the severity of both MR and TR, offering patients symptomatic relief and reductions in heart failure hospitalisation at low procedural risk. There is considerable geographic variation in protocols to assess these patients prior to the procedure and also in length of hospital stay. The standard of care in the UK, and particularly in Oxford, emphasises fewer investigations before the TEER procedure and shorter length of hospital stay.

This prospective, observational cohort study will examine the safety and feasibility of this practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Accepted by Heart Team for TEER (mitral and/or tricuspid)
* Willing and able to give informed consent for participation in the study.
* Regurgitation (mitral and/or tricuspid) grade ≥2+ as assessed by echocardiography
* Patient is willing and able to attend all follow-up visits

Exclusion Criteria:

* Patients in whom safety or clinical concerns preclude participation
* Patient declines to be involved in the study (unwilling to consent to enrolment or deemed by the patient advocate to be unwilling to consent)
* Patient in whom a TOE is contraindicated, or screening TOE is unsuccessful
* Pregnant or planning pregnancy within next 12 months
* Concurrent medical condition with a life expectancy of less than 12 months in the judgment of the Investigator
* Patients requiring emergency TEER

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged ≥18 years referred for either mitral or tricuspid TEER (or both) and found to be eligible candidates after review by the Oxford Heart Team.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients discharged 'early' after edge -to-edge repair | up to 30 days
  defined as < 36 hours after completion of procedure
All - cause rehospitalisation after completion of procedure | 30 days, 1 year
  Any hospital admission after discharge from the index procedure
All cause death after completion of procedure | 30 days, 1 year
  All patient death following discharge after the index procedure

SECONDARY OUTCOMES:
Hospital length of stay | Up to 3 months
  Length of hospital stay from admission to discharge for outpatient procedures, or from procedure to discharge for inpatient procedures
Proportion of patients requiring intensive care unit care | Up to 3 months
  The proportion of patients admitted to intensive care unit after their procedure
Safety outcomes a. Major adverse events at the time of the procedure b. Major adverse events (procedure/device related) up to 30 days | During index admission up to 30 days post procedure.
  Evaluating safety a. Major adverse events (procedure/device related) at the time of procedure b. Major adverse events (procedure/device related) up to 30 days (including unplanned surgery relating to a device/procedural complication)
Symptomatic improvement | 3 months, 1 year
  Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score from pre-procedure to post-procedure (validated score for assessing symptoms, physical and social limitations, and quality of life in patients with heart failure, score 0-100, where 100 = no symptoms).
Heart failure hospitalisation | 30 days, 1 year
  Any heart failure related hospitalisations after the index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Sam Dawkins, MBBS MRCP BSc DPhil, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No